CLINICAL TRIAL: NCT02387463
Title: Efficacy of Extended Peginterferon Alpha 2a(PEG-IFN a-2a) Treatment in HBeAg Positive Chronic Hepatitis B Patients
Brief Title: Efficacy of Extended Peginterferon Alpha 2a Treatment in HBeAg Positive Chronic Hepatitis B Patients
Status: Completed | Type: Observational
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, liver diseases center, Beijing Ditan Hospital
Other Study IDs: DTXY008
Record Dates: First submitted 2015-03-08; First posted 2015-03-13 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Chronic Hepatitis B
Keywords: chronic hepatitis B; antiviral therapy; peginterferon; HBeAg seroconversion; HBsAg loss
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The most important method to slow down and stop the liver disease progression in patients with chronic hepatitis B is antiviral therapy, by which to achieve maintaining viral response during treatment or obtain sustained viral response after treatment. The aim of the therapy with interferon is make patients obtain immune control to HBV, in clinical practice, it was expressed as HBeAg seroconversion, HBsAg loss and sustained viral response in HBeAg positive patients. However, those targets can't be get in most patients by 48 weeks of interferon treatment, and some patients need extended treatment to enhance the rate of HBeAg seroconversion and HBsAg loss. In this cohort study, the efficacies of extended therapy of interferon in HBeAg positive chronic hepatitis B patients will be evaluated.

DETAILED DESCRIPTION:
In this cohort study, the HBeAg positive chronic hepatitis B patients would be treated with peginterferon alpha 2a(PEG-IFN a-2a) for 96 week and followed 24 weeks after treatment. Serum HBV DNA load, HBsAg/anti-HBs level, HBeAg/anti-HBe will be tested at enrollment and every 3 months during treatment and follow period. Parameters of liver and kidney function, and liver ultrasound examination will be tested with intervals 1-3 months. The rates of HBeAg seroconversion, HBsAg loss, and sustained viral response will be evaluated after treatment and follow up.

ELIGIBILITY:
Inclusion Criteria:

* HBeAg positive chronic hepatitis B patients

Exclusion Criteria:

* Active consumption of alcohol and/or drugs
* Co-infection with human immunodeficiency virus, hepatitis C virus, or hepatitis D virus
* History of autoimmune hepatitis
* Psychiatric disease
* Evidence of neoplastic diseases of the liver

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: the population in this cohort study was composed of HBeAg positive chronic hepatitis B patients defined as HBsAg positive, HBeAg positive, and detectable HBV DNA load with ALT level ≥41 U/L for more than 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2012-03; Primary Completion 2017-05-21 (Actual); Study Completion 2017-05-21 (Actual)

PRIMARY OUTCOMES:
rate of HBeAg seroconversion (defined as HBeAg loss with anti-HBe positive after PEG-IFN a-2a treatment and follow up) | 120 weeks
  HBeAg seroconversion was defined as HBeAg loss with anti-HBe positive after PEG-IFN a-2a treatment and follow up.

SECONDARY OUTCOMES:
rate of HBsAg loss (defined as HBsAg level lower than 0.05 IU/ml) | 96 weeks
  HBsAg loss was defined as HBsAg level lower than 0.05 IU/ml.
rate of sustained viral response (defined as serum HBV DNA undetectable at the end of treatment and the end of follow up) | 120 weeks
  Sutained viral response was defined as serum HBV DNA undetectable at the end of treatment and the end of 24 weeks follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan hospital,Capital Medical University, Beijing, Beijing Municipality, China